CLINICAL TRIAL: NCT03483168
Title: The Effects of Culturally Sensitive Pain Education Program in Turkish Patients With Chronic Low Back Pain: A Pilot Randomized Controlled Trial
Brief Title: Culturally Sensitive Pain Education Program for Turkish Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceren Gürşen, Principal investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC UZG 2018/0228
Record Dates: First submitted 2018-03-16; First posted 2018-03-30 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally sensitive pain education (Experimental)
  Interventions: Behavioral: Culturally sensitive pain education
- Standard pain education (Active Comparator)
  Interventions: Behavioral: Standard pain education program

INTERVENTIONS:
Behavioral: Culturally sensitive pain education — The content of the PNE program include the characteristics of acute and chronic pain, purpose of acute pain, formation process of acute pain from the nervous system, the formation process of chronic pain, and potential sustaining factors for central sensitization.
  Arms: Culturally sensitive pain education
Behavioral: Standard pain education program — For the standard translated PNE, The English translation of "Pain Neuroscience Education: slides for supporting and illustrating your explanation" at the Pain in Motion Group web page (http://www.paininmotion.be/education/tools-for-clinical-practice) and English translation of the Patient Information Leaflet will be used. The education materials will be translated using the forward/backward translation process. The English version of PNE presentation and information leaflet will be translated to Turkish by two independent translators.
  Arms: Standard pain education

SUMMARY:
In last decade, the awareness has grown regarding the pain neuroscience education (PNE). In the literature, it has been found that there is strong evidence that the educational strategy of pain neuroscience education (PNE) can have positive effects on pain, disability, catastrophization, and physical performance in chronic musculoskeletal disorders. Nowadays, many physiotherapists integrate the PNE into the treatment of chronic pain. However, the importance of culturally sensitive approaches for the treatment of chronic pain has been proposed depending on the cultural differences of pain beliefs, pain cognitions, pain experiences and pain coping strategies in different ethnic populations. Therefore, the aim of this study is to compare the effects of a culturally sensitive PNE with a standard translated PNE on pain intensity, disability status, pain pressure thresholds and psychosocial factors (conceptualization of pain, pain beliefs, catastrophizing, kinesiophobia and illness perception) in Turkish patients with chronic low back pain (LBP).

The effects of culturally sensitive PNE format will be compared with the standard translated PNE in a pilot trial. 40 Turkish patients (first generation migrant living around Ghent) with chronic LBP, between the age of 18 and 65 years, will be randomized to the culturally sensitive PNE or standard translated PNE. The content of 2 sessions PNE include the explanation about differences of acute and chronic pain, purpose of acute pain, production of acute pain and chronic pain, and potential sustaining factors for central sensitization, but presented in different ways. They will be subjected to an individual education session and they will receive a home education program. In session 2 (after 1 week), they will come back to ascertain that everything is understood.

DETAILED DESCRIPTION:
In last decade, the awareness has grown regarding the pain neuroscience education (PNE). In the literature, it has been found that there is strong evidence that the educational strategy of pain neuroscience education (PNE) can have positive effects on pain, disability, catastrophization, and physical performance in chronic musculoskeletal disorders. Nowadays, many physiotherapists integrate the PNE into the treatment of chronic pain. However, the importance of culturally sensitive approaches for the treatment of chronic pain has been proposed depending on the cultural differences of pain beliefs, pain cognitions, pain experiences and pain coping strategies in different ethnic populations. Therefore, the aim of this study is to compare the effects of a culturally sensitive PNE with a standard translated PNE on pain intensity, disability status, pain pressure thresholds and psychosocial factors (conceptualization of pain, pain beliefs, catastrophizing, kinesiophobia and illness perception) in Turkish patients with chronic low back pain (LBP).

The effects of culturally sensitive PNE format will be compared with the standard translated PNE in a pilot trial. 40 Turkish patients (first generation migrant living around Ghent) with chronic LBP, between the age of 18 and 65 years, will be randomized to the culturally sensitive PNE or standard translated PNE. The content of 2 sessions PNE include the explanation about differences of acute and chronic pain, purpose of acute pain, production of acute pain and chronic pain, and potential sustaining factors for central sensitization, but presented in different ways. They will be subjected to an individual education session and they will receive a home education program. In session 2 (after 1 week), they will come back to ascertain that everything is understood.

The primary outcomes include pain intensity and disability status. Secondary outcome measures are pain pressure thresholds and psychosocial factors such as conceptualization of pain, pain Beliefs, catastrophizing, kinesiophobia and illness perceptions. Pain thresholds will be assessed with the pressure algometer. Pressure will be applied bilaterally at 3 pressure points: one on the mass of erector spinae muscle, one on the quadriceps muscle, and one on the trapezius muscle. All outcomes will be evaluated at baseline, day 7 (immediately after session 2) and after 1 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 40 Turkish patients between the age of 18 and 65 years, with a diagnosis of non-specific chronic LBP (have pain at least 3 months and mean pain frequency is 3 or more days per week), who are diagnosed by a physician and not starting new treatments,medication or continuing usual care 6 weeks prior and during study participation will be included to the present study. First generation Turkish migrants who are born in turkey, being Turkish as a first language, and being of Turkish nationality will be eligible for inclusion in this study.

Exclusion Criteria:

* Patients with uncontrolled mental health condition (eg, schizophrenia, bipolar disorder, major depressive disorder) that prevents the successful participation, specific pathologies, trauma, or pregnancy will be excluded. Study participants will be instructed to refrain from analgesics 48 hours prior to assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | change from baseline pain intensity at 4 week
  "0-10" Numerical Pain Scale
Disability status | Change from baseline disability status at 4 week
  Disability status will be assessed by using the Roland Morris Disability Questionnaire ranging from 0 to 24; higher scores represent higher levels of pain-related disability.

SECONDARY OUTCOMES:
Pain Pressure Thresholds | change from baseline pain pressure thresholds at 4 weeks
  Pain pressure thresholds will be assessed with a hand held pressure algometer (Wagner Force 50) with a circular probe of one cm diameter. Perpendicular pressure will be applied at a constant rate (1kg/s) to the tissue surface. 3 pressure-points will be evaluated bilaterally: One pressure points are on the Erector spinae muscle mass at 5 cm laterally of the processus spinosus vertebrae of L3, one pressure pain is on the middle of the quadriceps muscle (between the anterior superior iliac spine and base of the patella), one pressure point is on the middle of the trapezius muscle (between acromion and processus spinosus of C7). Two measurements will be taken with a 30 second interval and the mean of the measurements will be recorded.
Knowledge of pain | change from baseline pain knowledge at 4 weeks
  Knowledge of pain will be assessed by using the Revised Neurophysiology of Pain Questionnaire ranging from 0 to 13; higher scores represent higher levels of pain knowledge.
Pain related beliefs | change from baseline pain beliefs at 4 weeks
  Pain related beliefs will be assessed by using the Pain Beliefs Questionnaire consisting of two subscales: Organic Beliefs and Psychological Beliefs. Scores for each subscale ranges from 1 to 6; higher scores represent that having more negative pain beliefs.
Pain catastrophization | change from baseline pain catastrophization at 4 weeks
  Catastrophization of pain will be evaluated by using the Pain Catastrophizing Scale ranging from 0 to 52; higher scores represent higher levels of catastrophizing.
Fear avoidance beliefs related to pain | change from baseline kinesiophobia at 4 weeks
  Fear avoidance will be evaluated by using the Tampa Scale for Kinesiophobia ranging from 17 to 68; higher scores represent higher levels of kinesiophobia.
Illness perceptions | change from baseline illness perceptions at 4 weeks
  Illness perceptions will be evaluated by using the Brief Illness Perception Questionnaire; ranges from 0 to 80; higher scores represent a more threatening view of the illness.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Louw A, Puentedura EJ, Zimney K, Schmidt S. Know Pain, Know Gain? A Perspective on Pain Neuroscience Education in Physical Therapy. J Orthop Sports Phys Ther. 2016 Mar;46(3):131-4. doi: 10.2519/jospt.2016.0602. PMID 26928735
- [Result] Sleptsova M, Woessmer B, Grossman P, Langewitz W. Culturally sensitive group therapy for Turkish patients suffering from chronic pain: a randomised controlled intervention trial. Swiss Med Wkly. 2013 Nov 12;143:w13875. doi: 10.4414/smw.2013.13875. eCollection 2013. PMID 24222526
- [Result] Holzel LP, Ries Z, Kriston L, Dirmaier J, Zill JM, Rummel-Kluge C, Niebling W, Bermejo I, Harter M. Effects of culture-sensitive adaptation of patient information material on usefulness in migrants: a multicentre, blinded randomised controlled trial. BMJ Open. 2016 Nov 23;6(11):e012008. doi: 10.1136/bmjopen-2016-012008. PMID 27881523